CLINICAL TRIAL: NCT04024267
Title: Eurythmy Therapy (ERYT) as a Treatment Option for Fatigue in Metastatic Breast Cancer Patients
Acronym: ERYT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123123
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Fatigue; Breast Cancer
MeSH Terms: conditions — Fatigue; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eurythmy therapy (ERYT) (Experimental): Eurythmy therapy (ERYT) is a standardized movement therapy and for each medical condition standardized ERYT exercise (series) exist. In such, in the present study, the cancer series "O-E-M-L-I-B-D" that is specific and standardized for breast cancer patients will be applied. Patients can perform and maintain the postures without stress and tension. Patients are instructed by ERYT therapists in sessions with 1 to 4 patients.
  Interventions: Other: Eurythmy therapy
- CoordiFit (Active Comparator): The CoordiFit program consists of standardized exercises that address physical coordination, stability, balance and dexterity. These exercises serve as a control intervention and are non-specific with respect of cancer-related fatigue and breast cancer. They mimic those of ERYT but have no mindfulness features. Patients are instructed by physical therapists in session with 1 to 4 patients.
  Interventions: Other: CoordiFit

INTERVENTIONS:
Other: Eurythmy therapy — Mind-body therapy
  Arms: Eurythmy therapy (ERYT)
Other: CoordiFit — Fitness training
  Arms: CoordiFit

SUMMARY:
Cancer related fatigue (CRF) is the most burdening symptom in breast cancer patients, and prevalence exceeds 75% in patients with metastatic disease. CRF is described as the symptom that has the largest impact on quality of life, with negative effects on work, social activities, and daily activities, and may lead to treatment discontinuation. Currently, there is no gold standard for the treatment of CRF. Drug therapies are not satisfactory. Since physical activity is associated with significant reduction in CRF, patients are encouraged to engage in an at least moderate level of physical activity. However, for many metastatic breast cancer patients this is too burdensome. Finally, there is some evidence that non-pharmacological mind-body techniques may be beneficial in reducing CRF, yet the available data do not allow for final recommendations. Given the high prevalence of CRF and the substantial distress for patients, advancing treatment options for patients with CRF is highly desirable. In the present study, patients with metastatic breast cancer will be randomly assigned to two different non-pharmacological treatments for fatigue: Eurythmy therapy (ERYT), a standardized active mindful movement therapy, or a movement program without mindfulness features (CoordiFit). It will be tested, if ERYT has a superior benefit on fatigue compared to CoordiFit over the period of the intervention (20 weeks). Further, the benefit of ERYT on quality of life, sleep quality, anxiety, depression, pain, mobility of the arm, rate of return to work, compliance with ERYT, and targeted metabolomics will be investigated.

Both groups will have equal frequency and duration of the training sessions. Each patient will receive 13 standardized therapy sessions of 45 min (once a week for 6 weeks and once every second week) during the total period of 20 weeks. The proposed study has been developed in the Breast Cancer Project Group of the Swiss Group for Clinical Cancer Research (SAKK) and is supported by many breast centers, because they realize that the patients value non-pharmacological treatment options and would be keen to participate in such a trial. If ERYT proves to be beneficial, the impact of this trial will be high and will have implications not only for metastatic breast cancer patients but also for other cancer patients, health care personnel, scientists and funding and regulatory bodies.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 years or older
* Histologically or cytologically confirmed metastatic breast cancer
* FACIT-F subscale score < 34 (considered as cut-off for a diagnosis of relevant fatigue; a score < 30 is considered as severe fatigue [83])
* Eastern Cooperative Oncology Group (ECOG) grade 1 or 2
* Ability to physically and cognitively perform an active movement therapy
* Ability to provide informed consent as documented by signature
* Ability to read, write, and speak German, French, or Italian

Exclusion Criteria:

* Inability or contraindication that would prevent prolonged follow-up, or to undergo the investigated intervention or control intervention, in the opinion of the investigator
* Patients with psychiatric, addictive or any disorder that prevents the patient from adhering to the protocol requirements, in the opinion of the investigator
* Significant uncontrolled cardiac disease (e.g. unstable angina, recent myocardial infarction)
* Haemoglobin < 90 g/L

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fatigue over the whole intervention | End of the intervention (week 20)
  Fatigue is measured using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F). FACIT-F consists of the Functional Assessment of Cancer Therapy - General (FACT-G) plus the fatigue subscale comprising 13 fatigue-related items, with a total of 41 items. The fatigue subscale score is ranging from 8 to 44. A score < 34 is considered as cut-off for a diagnosis of relevant fatigue.

SECONDARY OUTCOMES:
Change from baseline in quality of life over the whole intervention | End of the intervention (week 20)
  Quality of life is measured using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F). FACIT-F consists of the Functional Assessment of Cancer Therapy - General (FACT-G) plus the fatigue subscale comprising 13 fatigue-related items, with a total of 41 items. The FACT-G subscale score ranges from 0 to 108. The higher the FACT-G subscale score the better the quality of life.
Change from baseline in patient's distress over the whole intervention | End of the intervention (week 20)
  Patient's distress is measured using the National Comprehensive Cancer Network (NCCN) Distress thermometer. The NCCN Distress thermometer ranges from 0 to 10, with 10 indicating an extreme distress and 0 indicating no distress.
Change from baseline in sleep quality over the whole intervention | End of the intervention (week 20)
  Sleep quality is measured using the Pittsburgh Sleep Quality Index (PSQI). The PSQI total score of the 9 items ranges from 0 to 21. A score < or = 5 is associated with good sleep quality; a score > 5 is associated with poor sleep quality.
Change from baseline in pain over the whole intervention | End of the intervention (week 20)
  Pain is measured using the Brief Pain Inventory (BPI). The BPI assesses pain at its "worst", "least", "average", and "now" (current pain). The four severity items range from 0 ("no pain") to 10 ("pain as bad as you can imagine").
Change from baseline in depression over the whole intervention | End of the intervention (week 20)
  Depression is assessed using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 total score for the nine items ranges from 0 to 27. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe, and severe depression, respectively.
Change from baseline in anxiety over the whole intervention | End of the intervention (week 20)
  Anxiety disorders are assessed using the General Anxiety Disorder-7 (GAD-7). The GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cutpoints for mild, moderate, and severe anxiety, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wolf, Professor, Study Chair — Institute for complementary and integrative medicine
Locations (11):
- Switzerland (11):
  - Brustzentrum Basel Bethesda Spital, Basel
  - St. Clara Forschung AG, Basel
  - Engeriedspital, Bern
  - University Hospital Bern, Bern
  - Institute of Complementary and Integrative Medicine, University of Bern, Bern
  - Hirslanden Bern AG, Salem-Spital, Brustzentrum Bern Biel, Bern
  - Tumorzentrum ZeTuP Rapperswil-Jona, Rapperswil-Jona
  - Tumor- und Brustzentrum ZeTuP AG, Sankt Gallen
  - Kantonsspital St.Gallen, Zentrum für Integrative Medizin, Sankt Gallen
  - Brustzentrum Ostschweiz AG, Sankt Gallen
  - Kantonsspital Winterthur, Medizinische Onkologie und Hämatologie, Winterthur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Timm E, Berlowitz I, Wolf U. Randomized controlled trial on eurythmy therapy versus slow-paced physical exercises for the treatment of fatigue in metastatic breast cancer patients. Oncologist. 2025 Nov 11;30(11):oyaf343. doi: 10.1093/oncolo/oyaf343. PMID 41123285
- [Derived] Meier-Girard D, Ribi K, Gerstenberg G, Ruhstaller T, Wolf U. Eurythmy therapy versus slow movement fitness in the treatment of fatigue in metastatic breast cancer patients: study protocol for a randomized controlled trial. Trials. 2020 Jul 6;21(1):612. doi: 10.1186/s13063-020-04542-5. PMID 32631427